CLINICAL TRIAL: NCT00759174
Title: Case Crossover Study of PDE5 Inhibitor Exposure as a Potential "Trigger Factor" for Acute NAION
Brief Title: A Study to Assess Whether PDE5 Inhibitors Increase the Chance of Triggering the Onset of Acute NAION
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481259
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Optic Neuropathy, Ischemic
Keywords: Optic Neuropathy Acute NAION PDE5 Inhibitor
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case Group
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention occurs in this observational study.

SUMMARY:
The objective of this non-interventional study is to examine whether use of Phosphodiesterase Inhibitors (PDE5s), including use of sildenafil, vardenafil, or tadalafil, triggers the onset of acute NAION.

DETAILED DESCRIPTION:
Sites will identify patients who meet the entry criteria during the conduct of their normal practice. Patients meeting these criteria will be offered participation in the study after reading and completing an informed consent document.

ELIGIBILITY:
Inclusion Criteria:

* Male aged ≥45 years;
* Experienced abrupt visual change in only 1 eye

Exclusion Criteria:

* Pain determined by an ophthalmologist to be consistent with an inflammatory/arteritic process or optic neuritis;
* History of NAION or optic neuritis.
* Participation in other studies within 60 days prior to entry in the study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential cases of acute NAION will be prospectively identified by approximately 125 ophthalmology centers in the US and Europe. Patients must have presented to an ophthalmologist within 3 weeks of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 673 (Actual)
Dates: Start 2008-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- United States (60):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Anchorage, Alaska
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Southbury, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Lisle, Illinois
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Lafayette, Louisiana
  - Pfizer Investigational Site, Ruston, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Beverly, Massachusetts
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, Chester, New Jersey
  - Pfizer Investigational Site, Newark, New Jersey
  - Pfizer Investigational Site, Roseland, New Jersey
  - Pfizer Investigational Site, Teaneck, New Jersey
  - Pfizer Investigational Site, Latham, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Woodbury, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- France (7):
  - Pfizer Investigational Site, Angers, Cedex 09
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Strasbourg
- Germany (10):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Tübingen
- Italy (7):
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Rome
  - Pfizer Investigational Site, Torino
- Spain (6):
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Cosalada
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Torrevieja
  - Pfizer Investigational Site, Valencia
- United Kingdom (3):
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Scarborough

REFERENCES:
- [Derived] Campbell UB, Walker AM, Gaffney M, Petronis KR, Creanga D, Quinn S, Klein BE, Laties AM, Lewis M, Sharlip ID, Kolitsopoulos F, Klee BJ, Mo J, Reynolds RF. Acute nonarteritic anterior ischemic optic neuropathy and exposure to phosphodiesterase type 5 inhibitors. J Sex Med. 2015 Jan;12(1):139-51. doi: 10.1111/jsm.12726. Epub 2014 Oct 31. PMID 25358826
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481259&StudyName=A%20Study%20to%20Assess%20Whether%20PDE5%20Inhibitors%20Increase%20the%20Chance%20of%20Triggering%20the%20Onset%20of%20Acute%20NAION

RESULTS

PARTICIPANT FLOW:
Groups:
- Potential NAION Cases With PDE5i Exposure: Participants who met pre-defined potential acute nonarteritic anterior ischemic optic neuropathy (NAION) criteria and were exposed to phosphodiesterase type 5 inhibitors (PDE5i) (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed.
- Potential NAION Cases Without PDE5i Exposure: Participants who met pre-defined potential acute NAION criteria and were not exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed.
Period: Overall Study
Arm/Group | Potential NAION Cases With PDE5i Exposure | Potential NAION Cases Without PDE5i Exposure
Started | 76 | 597
Completed | 76 | 595
Not Completed | 0 | 2
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Potential NAION Cases With PDE5i Exposure: Participants who met pre-defined potential acute NAION criteria and were exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed.
- Total: Total of all reporting groups
Arm/Group | Potential NAION Cases With PDE5i Exposure | Potential NAION Cases Without PDE5i Exposure | Total
Number analyzed (Participants) | 76 | 597 | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.3) | 62.3 (10.2) | 62.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 76 | 597 | 673

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Exposed to PDE5i During 1-Day Case Window and 29 1-Day Control Windows Among Participants Adjudicated as Definite NAION Cases
Description: Adjudication committee classified participants as Definite, Possible, or Non-NAION cases, or insufficient information available or unable to adjudicate. Case window: 1 day preceding symptom onset day; 29 control windows: 29 days preceding case window. A case or control window was considered exposed if: sildenafil/vardenafil was used on that day and/or previous day; tadalafil was used on that day and/or any of previous 4 days. In this analysis, each participant contributed exposure information for 1 case window and 29 control windows.
Time Frame: 30-day period prior to onset of NAION symptoms
Population: Full Analysis Set (FAS) included all participants who signed informed consent, were eligible for study, reported exposure to PDE5i within 60 days prior to participant-reported onset of NAION symptoms. N (number of participants analyzed) represents Definite NAION cases with PDE5i exposure on at least 1 day but not all 30 days prior to symptom onset.
Measure: Number; unit: exposed days
Units Other Than Participants: Days
Groups:
- Potential NAION Cases With PDE5i Exposure/ Case Window: Participants who met pre-defined potential acute NAION criteria and were exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed. Case window is the day preceding the symptom onset day.
- Potential NAION Cases With PDE5i Exposure/ Control Window: Participants who met pre-defined potential acute NAION criteria and were exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed. Control windows are the 29 days preceding the case window.
Arm/Group | Potential NAION Cases With PDE5i Exposure/ Case Window | Potential NAION Cases With PDE5i Exposure/ Control Window
Number analyzed (Participants) | 43 | 43
Number analyzed (Days) | 43 | 1247
exposed days | 14 | 248
Statistical Analysis 1: Comparison: Potential NAION Cases With PDE5i Exposure/ Case Window vs Potential NAION Cases With PDE5i Exposure/ Control Window; Conditional logistic regression was stratified by participant; Test type: Superiority or Other; p = 0.033, Conditional logistic regression; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.06 to 4.34]

2. Other Pre Specified Outcome: Number of Days Exposed to PDE5i During 1-Day Case Window and 29 1-Day Control Windows Among Participants Adjudicated as Definite or Possible NAION Cases
Description: as for outcome 1
Time Frame: 30-day period prior to onset of NAION symptoms
Population: FAS included all participants who signed informed consent, were eligible for study and reported exposure to PDEi within 60 days prior to participant reported-onset of NAION symptoms. N (number of participants analyzed) represents Definite or Possible NAION cases with PDE5i exposure on at least 1 day but not all 30 days prior to symptom onset.
Measure: Number; unit: exposed days
Units Other Than Participants: Days
Arm/Group | Potential NAION Cases With PDE5i Exposure/ Case Window | Potential NAION Cases With PDE5i Exposure/ Control Window
Number analyzed (Participants) | 64 | 64
Number analyzed (Days) | 64 | 1856
exposed days | 22 | 374
Statistical Analysis 1: Comparison: Potential NAION Cases With PDE5i Exposure/ Case Window vs Potential NAION Cases With PDE5i Exposure/ Control Window; Conditional logistic regression was stratified by participant; Test type: Superiority or Other; p = 0.003, Conditional logistic regression; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.33 to 4.19]

3. Other Pre Specified Outcome: Number of Weeks Exposed to PDE5i During 1-Week Case Window and 7 1-Week Control Windows Among Participants Adjudicated as Definite NAION Cases
Description: Adjudication Committee classified participants as Definite, Possible, or Non-NAION cases, or insufficient information available or unable to adjudicate. Case window: 1 week preceding symptom onset day; 7 control windows: 7 weeks preceding case window. 1-week case or control window was considered exposed if any of 7 days were classified as exposed (sildenafil/vardenafil used on given day and/or previous day, or tadalafil used on given day and/or previous 4 days). In this analysis, each participant contributed exposure information for 1 case window and 7 control windows.
Time Frame: 60-day period prior to onset of NAION symptoms
Population: FAS population. N (number of participants analyzed) represents Definite NAION cases with PDE5i exposure on at least 1 day but not all 30 days or every week within 60 days prior to symptom onset.
Measure: Number; unit: exposed weeks
Units Other Than Participants: Weeks
Groups:
- Potential NAION Cases With PDE5i Exposure/ Case Window: Participants who met pre-defined potential acute NAION criteria and were exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed. Case window is the week preceding the symptom onset day.
- Potential NAION Cases With PDE5i Exposure/ Control Window: Participants who met pre-defined potential acute NAION criteria and were exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed. Control windows are the 7 weeks preceding the case window.
Arm/Group | Potential NAION Cases With PDE5i Exposure/ Case Window | Potential NAION Cases With PDE5i Exposure/ Control Window
Number analyzed (Participants) | 36 | 36
Number analyzed (Weeks) | 36 | 252
exposed weeks | 23 | 91
Statistical Analysis 1: Comparison: Potential NAION Cases With PDE5i Exposure/ Case Window vs Potential NAION Cases With PDE5i Exposure/ Control Window; Conditional logistic regression was stratified by participant; Test type: Superiority or Other; p < 0.001, Conditional logistic regression; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.70 to 7.69]

ADVERSE EVENTS:
Description: Given retrospective data collection, adverse events may have occurred prior to informed consent.
Groups:
- Potential NAION Cases: All participants who met pre-defined potential acute NAION criteria and were either exposed or not exposed to PDE5i (sildenafil, vardenafil or tadalafil) during the 60 days prior to NAION symptom onset were observed.
Arm/Group | Potential NAION Cases
Serious Adverse Events (participants affected / at risk) | 2/673
Other Adverse Events (participants affected / at risk) | 0/673
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Potential NAION Cases (N=673)
Diarrhoea (Gastrointestinal disorders) | 1
Candidiasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Blood pressure decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Haemorrhage (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Potential for bias from inaccuracies in recall of exposure and exposure-based enrollment were evaluated. Although these sources of bias cannot be excluded, they were unlikely to have substantially affected the primary results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.